CLINICAL TRIAL: NCT03976609
Title: Three Dimensional Changes on Nasal Septum and Alveolar Cleft After Maxillary Expansion: A Case Series
Brief Title: Three Dimensional Changes on Nasal Septum and Alveolar Cleft After Maxillary Expansion
Status: Completed | Type: Observational
Sponsor: Pontifícia Universidade Católica de Minas Gerais (Other)
Responsible Party: Principal Investigator, Ildeu Andrade Jr., Associate Professor, Pontifícia Universidade Católica de Minas Gerais
Other Study IDs: Maxillary Expansion Cleft Pts
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Nasal Septum; Deviation, Congenital; Cleft Lip and Palate; Maxillary Hypoplasia
Keywords: Nasak Septum; Cleft Lip; Cleft palate; Palatal expansion technique
MeSH Terms: conditions — Cleft Lip; Retrognathia; Cleft Palate | interventions — Palatal Expansion Technique

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Maxillary Expansion — The patients with maxillary transverse deficiency were treated with Haas expander is a tooth and tissue-borne appliance with a jackscrew located at the anterior region of the arch with its arms bent posteriorly and soldered to the first permanent molar bands. Once activated, the appliances opens the palatal suture and increase the transverse dimension of the maxilla.
  Other Names: Palatal expansion technique

SUMMARY:
This study evaluates, by means of cone beam computed tomography (CBCT), the alterations in the nasal septum and alveolar cleft volume that occur in cleft lip and palate (CLP) patients after rapid maxillary expansion(RME). 40 unilateral CLP patients (mean age, 11.1 ± 2.2 years) with transverse maxillary deficiency that underwent to RME will be evaluated in this investigation. CBCT images were taken prior to RME (T0) and after the removal of the expander (T1), for adequate secondary bone graft surgical planning. The scans will be used to analyze the effects on the nasal septum, anterior and posterior maxillary basal width (MBW) and alveolar cleft volume.

DETAILED DESCRIPTION:
Rapid maxillary expansion (RME) is performed to correct crossbite in CLP patients as part of the orthodontic treatment, being able to improve the maxillary transverse dimension, that is an essential condition for alveolar bone grafting. The primary aim of the secondary graft surgery is to restore the function and structure of the maxillary arch at the cleft side, providing support to arch width, minimizing its transverse collapse. However, since RME exert heavy forces to separate the two maxillary helves, it may significantly widen the alveolar cleft defect, possibly compromising bone graft success.

Moreover, RME has an important impact on the geometry and function of the nasal cavity, providing a lateral displacement of the walls and facilitating the airflow through the upper airways. These effects are very important to CLP patients, since they usually present reduced upper airway dimensions, adenoid hypertrophy, sleep disorders, oral breathing, and a marked nasal septal deviation. The nasal septal deviation is one of the major causes of nasal obstruction in non-cleft patients, and often results in blocking of the nasolacrimal ducts, sinusitis, ear infections and mouth breathing. However, nasal septum deviation in CLP patients commonly persists even after surgical repair of the cleft, leading to a chronic obstruction of the air passage, until the septorhinoplasty, at the age of 14-18 years.

Each expander was cemented with a fluoride releasing cement, and the activation regimen was established at 2 turns/day until the tip of the lingual cusps of the maxillary teeth touched the tips of the buccal cusps of the mandibular teeth. After the 3-month retention period, the expander was removed, and a post-expansion CBCT scanning (T1) was acquired for adequate secondary bone graft surgical planning.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria comprehended the presence of unilateral cleft lip and palate, rapid maxillary expansion as an initial part of the orthodontic treatment, and absence of previous orthodontic treatment.

Exclusion Criteria:

* The exclusion criteria were absent maxillary permanent first molars, signs of active periodontal disease, and presence of any additional craniofacial syndrome.

Ages: 8 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: 40 unilateral cleft lip and palate patients (UCLP) (23 male and 17 female), aging from 8 to 14 years old (mean age of 11.1 years ± 2.2). All subjects were in prepubertal or pubertal stage of maturation based on the cervical vertebrae maturation19 assessed on reconstructed lateral cephalograms generated from CBCT.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Alterations on Nasal septum | 1 - 2 months
  Maxillary expansion performed with 2 activations per day until the tip of the lingual cusps of the maxillary teeth touched the tips of the buccal cusps of the mandibular teeth.
Changes in the alveolar cleft dimensions | 1 - 2 months
  Maxillary expansion performed with 2 activations per day until the tip of the lingual cusps of the maxillary teeth touched the tips of the buccal cusps of the mandibular teeth.

SECONDARY OUTCOMES:
Anterior and posterior maxillary basal width changes | 1 - 2 months
  Maxillary expansion performed with 2 activations per day until the tip of the lingual cusps of the maxillary teeth touched the tips of the buccal cusps of the mandibular teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Ildeu Andrade Jr., DDS, MS, PhD, Principal Investigator — Pontifícia Universidade Católica de Minas Gerais

IPD SHARING:
Plan to Share IPD: No
Patient's individual data might be available upon a reasonable request

REFERENCES:
- [Background] Jiang M, You M, Wang S, Wang K, Feng B, Wang H. Analysis of Nasal Septal Deviation in Cleft Palate and/or Alveolus Patients Using Cone-Beam Computed Tomography. Otolaryngol Head Neck Surg. 2014 Aug;151(2):226-31. doi: 10.1177/0194599814531022. Epub 2014 Apr 16. PMID 24740983
- [Background] Aziz T, Wheatley FC, Ansari K, Lagravere M, Major M, Flores-Mir C. Nasal septum changes in adolescent patients treated with rapid maxillary expansion. Dental Press J Orthod. 2016 Jan-Feb;21(1):47-53. doi: 10.1590/2177-6709.21.1.047-053.oar. PMID 27007761
- [Background] Mordente CM, Palomo JM, Horta MC, Souki BQ, Oliveira DD, Andrade I Jr. Upper airway assessment using four different maxillary expanders in cleft patients: A cone-beam computed tomography study. Angle Orthod. 2016 Jul;86(4):617-24. doi: 10.2319/032015-174.1. Epub 2015 Nov 23. PMID 26595658
- [Background] Quereshy FA, Barnum G, Demko C, Horan M, Palomo JM, Baur DA, Jannuzzi J. Use of cone beam computed tomography to volumetrically assess alveolar cleft defects--preliminary results. J Oral Maxillofac Surg. 2012 Jan;70(1):188-91. doi: 10.1016/j.joms.2011.01.027. Epub 2011 May 6. PMID 21549490
- [Background] Long RE Jr, Spangler BE, Yow M. Cleft width and secondary alveolar bone graft success. Cleft Palate Craniofac J. 1995 Sep;32(5):420-7. doi: 10.1597/1545-1569_1995_032_0420_cwasab_2.3.co_2. PMID 7578207